CLINICAL TRIAL: NCT06933771
Title: The Effectiveness of Lavender Essence in Reducing Pain and Fear in Children During Blood Draws; A Randomized Controlled Study
Brief Title: Children's Blood Draws: Lavender Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corlu State Hospital (Other Government)
Responsible Party: Principal Investigator, Gülsev Kutman, Nurse, Corlu State Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Çorlu State Hospital
Record Dates: First submitted 2023-10-27; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Nursing Caries; Pain Management
Keywords: PAİN; FEAR
MeSH Terms: conditions — Agnosia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: LAVENDER ESSENCE GROUP - CONTROL GROUP
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LAVENDER ESSENCE GROUP (Active Comparator): the researcher explained to the children in the intervention group and their parents how to apply the lavender essence and what kind of a plant lavender is, and showed the bottle of essential oil to be used during the procedure. A 5x5 cm sponge with 2 drops of almond oil that contains 1% lavender essence was located on the shoulder of the children to smell for 5 minutes.
  Interventions: Other: LAVENDER ESSENCE GROUP
- CONTROL GROUP (Sham Comparator): no intervention was made.
  Interventions: Other: CONTROL GROUP

INTERVENTIONS:
Other: LAVENDER ESSENCE GROUP — Parents stood on the left side, easily visible to the child. The sole routine method used to reduce pain in the blood collection unit of the hospital in which the study was conducted is the presence of parents during the procedure. In this study, all children in both intervention and control groups were accompanied by their parents. Afterwards, the researcher explained to the children in the intervention group and their parents how to apply the lavender essence and what kind of a plant lavender is, and showed the bottle of essential oil to be used during the procedure. A 5x5 cm sponge with 2 drops of almond oil that contains 1% lavender essence was located on the shoulder of the children to smell for 5 minutes.
  Other Names: AROMATHERAPY GROUP
  Arms: LAVENDER ESSENCE GROUP
Other: CONTROL GROUP — Parents stood on the left side, easily visible to the child. The sole routine method used to reduce pain in the blood collection unit of the hospital in which the study was conducted is the presence of parents during the procedure. In this study, all children in both intervention and control groups were accompanied by their parents. Routine nursıng care provıed.
  Arms: CONTROL GROUP

SUMMARY:
The aim of this study is to show the effect of lavender scent used to reduce pain and fear during blood collection in children aged 7-14.

DETAILED DESCRIPTION:
The children in the experimental group were given lavender scent before the blood collection procedure. No additional intervention was made to the children in the control group. The pain and fear scores of both groups were evaluated.

ELIGIBILITY:
Inclusion Criteria:

children between the ages of 7-14 who applied to the blood collection unit, who had no mental neurological, hearing, speech, vison disorders

Exclusion Criteria:

who were not allergic to lavender essence, who were not diagnosed with asthma, allergies, epilepsy, dermatitis who had not taken analgesics in the last 6 hours were included in the study

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Child Medical Fear Scale (CMFS) | 9 MONTHS
  It is a 3-point Likert type scale that includes 29 items expressing the medical fears of children. For each item, the child is asked to choose one of the following responses: "not all afraid" (1), "a little afraid" (2), "very afraid" (3). The scale has 4 subscale dimensions which are procedural fears, environmental fears, intrapersonal fears and interpersonal fears. The total score that can be obtained on the scale ranges from 29 as the lowest to 87 as the highest .
  Children who score between 0-29 points are considered "not afraid" while the children who score between 29-58 points are considered "a little afraid", and children who score between 58-87 points are considered "very afraid".
Wong-Baker FACES Pain Rating Scale (WBFPRS) | 9 MONTHS
  On the scale, there are 6 facial expressions that are presented on a horizontal plane and scored from 0 to 10. The happy facial expression on the far left represents a score of 0, meaning "doesn't hurt at all" and the crying facial expression on the far right represents a score of 10, meaning "hurts as much as you can imagine

CONTACTS AND LOCATIONS:
Locations (1):
- Çorlu State Hospital, Merkez, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No